CLINICAL TRIAL: NCT03063918
Title: Pilot Study of a Personalized Dietary Intervention to Manage Bowel Dysfunction in Rectal Cancer Survivors
Brief Title: Personalized Dietary Intervention in Managing Bowel Dysfunction and Improving Quality of Life in Stage I-III Rectosigmoid Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Hope Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16332; NCI-2017-00258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16332 (Other: City of Hope Medical Center)
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Cancer Survivor; Stage I Rectosigmoid Cancer; Stage II Rectosigmoid Cancer; Stage III Rectosigmoid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (personalized dietary intervention) (Experimental): At 6 months after standard of care treatment, patients receive 10 sessions of personalized dietary intervention over 30 minutes each over 4 months via the telephone. Patients also receive a workbook including reference materials and intervention content.
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Informational Intervention — Receive a workbook
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive personalized dietary intervention

SUMMARY:
This pilot clinical trial studies how well personalized dietary intervention works in managing bowel dysfunction and improving quality of life in stage I-III rectosigmoid cancer survivors. Personalized dietary intervention may help people understand bowel symptoms, identify helpful and troublesome foods for bowel symptoms, adjust diets and food preparation based on food triggers, and coach on healthy diet recommendations after cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Administer and determine the feasibility of the personalized dietary intervention.

II. Using qualitative methods, evaluate the acceptability of the intervention as reported by survivors.

III. Explore decisional conflict associated with treatment decision-making in rectal cancer surgery.

OUTLINE:

At 6 months after standard of care treatment, patients receive 10 sessions of personalized dietary intervention over 30 minutes each over 4 months via the telephone. Patients also receive a workbook including reference materials and intervention content.

After completion of study, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-III cancers of the rectosigmoid colon or rectum
* 6 months post-treatment completion
* Have a permanent ostomy or anastomosis
* English-speaking
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with stage IV disease will be excluded from the study
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Acceptability assessed by semi-structured interview | Up to 6 months
  Will be assessed through qualitative data analysis using conventional content analysis approach.
Bowel function assessed by Memorial Sloan Kettering Cancer Center Bowel Function Tool | Up to 6 months
  Descriptive statistics will be summarized using validated scoring procedures.
Feasibility assessed by patient enrollment | Up to 6 months
  Will be assessed through: 1) the ratio of eligible participants to those enrolled and those who declines participation; 2) reasons for non-participation; 3) number of scheduled study encounters completed; 4) attrition rate between pre- and post-intervention; 5) reasons for attrition/dropout; 6) level of intervention participation including the total number of sessions, number of sessions completed without break-offs, number of break-offs, length (minutes) of sessions; and 7) the ratio of all participants to those who complete >= 80% of the study.
Quality of life assessed by City of Hope-Quality of Life-Colorectal Cancer | Up to 6 months
  Descriptive statistics will be summarized using validated scoring procedures.

OTHER OUTCOMES:
Scores from the Decisional Conflict Scale | Up to 6 months
  Descriptive statistics will be summarized. This analysis is exploratory only. Will use the findings to support future research related to treatment-decision making in rectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, PhD, RN, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - City of Hope Medical Center, Duarte, California